CLINICAL TRIAL: NCT06143423
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial to Evaluate AP026 (TQA2226) for Injection in Adult Subjects After Single/Multiple Administration.
Brief Title: A Clinical Trial of AP026 (TQA2226) for Injection in Adult Subjects.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQA2226-I-01
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AP026 (TQA2226) for injection Single administration dose (SAD) (Experimental): AP026 (TQA2226) for injection, administered once.
  Interventions: Drug: AP026 (TQA2226) for injection
- AP026 (TQA2226) for injection matching placebo Single administration dose (SAD) (Placebo Comparator): AP026 (TQA2226) for injection matching placebo, administered once.
  Interventions: Drug: AP026 (TQA2226) for injection matching placebo
- AP026 (TQA2226) for injection Multiple administration dose (MAD) (Experimental): AP026 (TQA2226) for injection, administered 4 times.
  Interventions: Drug: AP026 (TQA2226) for injection
- AP026 (TQA2226) for injection matching placebo Multiple administration dose (MAD) (Placebo Comparator): AP026 (TQA2226) for injection matching placebo, administered 4 times.
  Interventions: Drug: AP026 (TQA2226) for injection matching placebo

INTERVENTIONS:
Drug: AP026 (TQA2226) for injection — AP026 (TQA2226) for injection is a GLP-1-FGF21-Fc bifunctional fusion protein.
  Arms: AP026 (TQA2226) for injection Multiple administration dose (MAD); AP026 (TQA2226) for injection Single administration dose (SAD)
Drug: AP026 (TQA2226) for injection matching placebo — AP026 (TQA2226) for injection matching placebo is a placebo produced according to AP026 (TQA2226) for injection, and has no effect on GLP-1 and FGF21.
  Arms: AP026 (TQA2226) for injection matching placebo Multiple administration dose (MAD); AP026 (TQA2226) for injection matching placebo Single administration dose (SAD)

SUMMARY:
This study was a randomized, double-blind, placebo-controlled phase I clinical trial of AP026 (TQA2226) for injection in adult healthy subjects, which planned to recruit 74 healthy subjects. The main purpose was to evaluate the safety and tolerance of AP026 (TQA2226) for injection after single and multiple doses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Sign an informed consent form before the study and have a thorough understanding of the content, process, and potential adverse reactions of the study;
* Able to complete the study according to the requirements of the protocol;
* Subjects (including their partners) are willing to voluntarily take effective contraceptive measures within 6 months after the last study drug administration;
* Male and female subjects aged 18-55 (inclusive);
* Male subjects weighing no less than 50 kilograms and female subjects weighing no less than 45 kilograms, With a body mass index within the range of 18~28kg/m2 (inclusive);
* Physical examination and vital signs are normal or abnormal but with no clinical significance (judged by the investigators).

Exclusion Criteria:

* Pregnant and lactating women;
* There are abnormal and clinically significant clinical laboratory examination results, or clinically significant diseases within 12 months before screening, which is not recommended to participate in the trial after evaluation by the investigators. Subjects with a previous medical history but are recovered with clinical evidence can be included in this study;
* During the screening period, any one of the vital signs, physical examination, laboratory examination, 12 lead electrocardiogram, and other auxiliary examination results is abnormal and judged by the investigator to have clinical significance;
* Subjects who test positive for any of the hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (Anti HCV), human immunodeficiency virus antibody (Anti HIV), and Treponema pallidum antibody (Anti TP);
* Those who have undergone surgery within 4 weeks before screening or plan to undergo surgery during the study period;
* Received investigational drugs or participated in clinical trials within 3 months prior to screening;
* Received immunoglobulin or blood products within 30 days before randomization;
* Donated blood (> 300 mL) or experienced significant blood loss (> 400 mL) within 3 months prior to screening;
* Subjects with a history of needle sickness, blood sickness, or potential difficult in collecting blood;
* History of allergic reactions to other therapeutic monoclonal antibodies or biological agents, or history of allergies to multiple drugs or foods, especially to ingredients similar to the study drug;
* Smoking more than 5 cigarettes per day or using an equivalent amount of nicotine or nicotine containing products within 3 months before randomization, or failing to stop using any tobacco products during the trial period;
* Those who have been drinking excessively for a long time or have consumed more than 14 units of alcohol per week within 3 months before screening, or cannot abstain from alcohol during the trial period, or have tested positive for alcohol breath test;
* Subjects with a history of drug abuse, or positive urine drug screening;
* Received any commercially available or investigational biological agents within 4 months before randomization or within 5 half-lives of drugs (whichever is longer);
* Within 4 weeks before randomization, received any systemic prescription drugs, over-the-counter drugs, herbs, any vitamin products, and health products, or any topical drugs of the above forms at the injection site of this study;
* From the screening period to the study medication, acute diseases or concomitant medication occured.
* Any medical history that may affect drug absorption, distribution, metabolism, and excretion.
* Any situation that the investigator believes will pose a safety risk to the subject during the study or may interfere with the implementation of this study, or the investigator believes that the subject may not be able to complete this study or may not be able to comply with the requirements of this study.
* QT interval > 450 milliseconds, or electrocardiogram is not suitable for Concentration-QT measurement (according to the judgment of the investigator).
* History of risk factors for torsade de pointe ventricular tachycardia. Subject with a family history of long QT syndrome or Brugada syndrome will also be excluded.
* Heart rate ≤ 45 bpm.
* History of renal or liver dysfunction.
* History or condition of cardiovascular disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From patient enrollment to withdrawal, estimated up to 2 months.
  Incidence of adverse events after dose, assessed by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
Severity of adverse events | From patient enrollment to withdrawal, estimated up to 2 months.
  Severity of adverse events after dose, assessed by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
Incidence of serious adverse events (SAEs) | From patient enrollment to withdrawal, estimated up to 2 months.
  Incidence of serious adverse events after dose, assessed by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
Severity of serious adverse events (SAEs) | From patient enrollment to withdrawal, estimated up to 2 months.
  Severity of serious adverse events after dose, assessed by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.

SECONDARY OUTCOMES:
Peak concentration (Cmax) | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  The highest blood drug concentration achieved after administration.
Plasma concentration-area under time curve (AUC0-t) | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  The area under the plasma concentration-time curve from the beginning of the first administration to the last measurable concentration point.
Plasma concentration-area under time curve (AUC0-∞) | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  Extrapolated from the first administration to the area under the plasma concentration-time curve to infinity.
Peak Time (Tmax) | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  the time required to reach the highest concentration (peak drug concentration).
Apparent volume of distribution (Vd/F) | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  The theoretical volume that would be necessary to contain the total amount of an administered drug at the same concentration that it is observed in the blood plasma
Clearance (CL) | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  The volume of a substance in plasma that the body or organ can clear per unit time.
Elimination half-life time (t1/2) | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  The time it takes to reduce the concentration of drugs in the blood by half.
Plasma concentration at steady state (Cav, SS) | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  The plasma concentration at which the rate of administration and rate of elimination are in equilibrium.
Tmax, ss | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  Time required to reach steady-state peak concentration after administration
Cmax, ss | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  The highest blood drug concentration that occurs after reaching steady state
Cmin, ss | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  The lowest blood drug concentration that occurs after reaching steady state
AUC, ss | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  The area under the plasma concentration-time curve of the steady state
Rac | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  The ratio of steady-state blood drug concentration to blood drug concentration after the first administration
Anti-Drug Antibody (ADA) | SAD: From 30 minutes before administration to 1176 hours after administration on Day 1. MAD: From 30 minutes before administration on Day 1 to 1008 hours after the last administration.
  The incidence of ADA after drug administration for evaluating the immunogenicity of antibody drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China